CLINICAL TRIAL: NCT04055350
Title: Electronically Recorded National Early Warning Scores, Pain Scores and PONV Scores Among Hospitalized Patients and the Associated Patient Outcomes.
Brief Title: Electronically Recorded National Early Warning Scores, Pain Scores and PONV Scores Among Hospitalized Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Joonas Tirkkonen, MD, PhD. Resident in Anaesthesiology and Intensive Care Medicine. Principal Investigator in this Study., Tampere University Hospital
Other Study IDs: R20007R
Record Dates: First submitted 2019-08-05; First posted 2019-08-13 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Prevention of In-hospital Adverse Events
Keywords: National early warning score; Prevention of serious adverse events; Patient deterioration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
National early warning score (NEWS) enables early detection of patient deterioration in hospital floors. However, there is limited data on the prognostic value of NEWS among actual general ward patients. Further, there is no data on how changes in NEWS-values impact patient outcomes. Very little is known on how post-operative nausea and vomiting (PONV) and pain influences NEWS values and vital signs in general.

DETAILED DESCRIPTION:
The investigators aim to collect detailed data on patients' vital signs, NEWSs, pain scores and PONV scores through electronic data records, where these values are automatically stored with mobile mobile smart devices used by nursing staff. The expected volume of the cohort is 50,000 patients and 300,000 recordings of vital signs.

In addition to the scores and vital signs, the registry will include patients' identification numbers (IDs), dates and times of the recordings, and ward numbers. With the IDs, mortality data up to 90-days for the patients will be obtained from the national population register centre. All data will be handled in a pseudonymized form in a secure computer inside hospital, and approval to use the registry in study purposes will be obtained from the Ethics Committee of Tampere University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Adult in-hospital patients with recordings of vital signs

Exclusion Criteria:

* Patients under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult in-hospital patients in Pirkanmaa Hospital District whose vital signs have been recorded with mobile smart devices during the study period.
Sampling Method: Probability Sample
Enrollment: 30000 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Death occurring within 90-days of the last NEWS measurement | 90 days
  The percentage of patients that die within 90-days of the last NEWS recording during their hospitalization.
Death occurring within one day after the first NEWS measurement on general wards | One day
  The percentage of patients that die within one day after their first NEWS measurement at the beginning of their general ward admission

SECONDARY OUTCOMES:
Death occurring within 30-days of the last NEWS measurement | 30 days
  The percentage of patients that die within 30-days of the last NEWS recording during their hospitalization.
Death occurring within 2-30 days after the first NEWS measurement on general wards | 2-30 days
  The percentage of patients that die within 2-30 days after their first NEWS measurement at the beginning of their general ward admission
Incidence of post operative nausea and vomiting | Up to 30 days after the first recording of patient's vital signs in the electronic patient records
  Percentage of patients suffering from post-operative nausea and vomiting (recorded as a scale from 0 to 5) in the electronic patient records.
Incidence of post operative pain | Up to 30 days after the first recording of patient's vital signs in the electronic patient records
  Percentage of patients suffering from post operative pain (recorded as numerical scale from 0 to 10) in the electronic patient records.

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital, Tampere, Pirkanmaa, Finland

IPD SHARING:
Plan to Share IPD: No
Due to data security policies, individual participant data will not be shared.

REFERENCES:
- [Derived] Loisa E, Kallonen A, Hoppu S, Tirkkonen J. Ability of the National Early Warning Score and its respiratory and haemodynamic subcomponents to predict short-term mortality on general wards: a prospective three-centre observational study in Finland. BMJ Open. 2022 Apr 26;12(4):e055752. doi: 10.1136/bmjopen-2021-055752. PMID 35473725